CLINICAL TRIAL: NCT04441853
Title: Use of YouTube as a Teaching Tool for Nursing Student to Learn About Empathy
Brief Title: Use of YouTube for Nursing Students to Learn Empathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tung Wah College (Other)
Responsible Party: Principal Investigator, Siu Mei Yi, Principal Investigator, Tung Wah College
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RESC2018001
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2020-06-24 (Actual); Status verified 2020-06

CONDITIONS: Nurse-Patient Relations
Keywords: YouTube; teaching; nursing student; emapthy

STUDY DESIGN:
Intervention Model Description: The convenience samples were two groups of students enrolled in a geriatric nursing course at two consecutive semesters, from the school of nursing, in a tertiary education institution in Hong Kong. Students who studying the geriatric course in the first semester were treated as intervention group, whereas students studying the same course in the second semester were assigned as control.
  Students of the intervention group were invited to view a series of YouTube video, comprising five sessions, related to geriatric course content and focusing on patients' and caregivers' lived experience. Then, they were requested to participate in group discussion to stimulate their learning and understanding of patients' and caregivers' situation. Meanwhile, students of the control group were taught with the same content through the usual lecture-based method, without You Tube video.
Masking Description: All personals involved the study (students, teachers, investigators and outcome assessors) had not been masked for treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YouTube video group (Experimental): The intervention group attended five sessions of weekly-based tutorial, by watching YouTube videos on older people's and their caregivers' lived experience. On each session, they would joined post-video group discussion.
  Interventions: Other: YouTube video
- No YouTube video group (Active Comparator): The control group were offered for five sessions of tutorial with same content without YouTube or other audio-visual tools. They also needed to join for group discussion in each tutorial.
  Interventions: Other: Control

INTERVENTIONS:
Other: YouTube video — Tutoral session on using YouTube personal stories on older people
  Arms: YouTube video group
Other: Control — Tutorial session with same content without Youtube video
  Arms: No YouTube video group

SUMMARY:
Caring is an integral part of nursing. It is grounded on universal human value such as empathy, to provide quality nursing care to patients. Nursing educators have a responsibility to develop teaching strategies to enable students to learn how to care using empathy. One way to foster empathy is by adopting experiential learning where knowledge and understanding is developing through transforming of experience. The use of cinema, as a form of drama, provides opportunities for students to learn from another people's story. You Tube, a large medium of digital story video clips, can offers tremendous opportunities for nursing educators to engage and assess to students. Some You Tube videos provide fictional scenarios from people discussing on their health problems and related concerns that give students real-life insight and promote cultivation on empathetic caring attitudes required for ethical healthcare practice needs. Using video technology to facilitate learning has become more popular in nursing but the research for using YouTube as a pedagogical tool on empathy is limited.

This study aims to examine the use of YouTube video as a teaching resource on nursing student's empathy, attitude and understanding of patients' and caregivers' experience in various health conditions.

DETAILED DESCRIPTION:
1. Study design, sampling and data collection This study is a mixed study design, using questionnaires and focus group discussions for data collection. The study period involves two semesters for the academic year. A convenience non-probability sampling method will be employed.

   The first part of the study is planned for quantitative data collecting, it adopts a quasi-experimental, non-equivalent pre- and post-control group design. Both group of students are recruited from two different semesters who study for the same geriatric course. Students enroll for the geriatric course in the first semester are treated as the intervention group, while students study the same course in next semester are assigned for the control group. Both groups are assessed by the pre- and post-test to investigate on change of students' empathy by the Taiwan version of Jefferson Scale of Empathy - Health Professions Students (C-JSE-HPS). Additionally, students of the intervention group will be assessed on their perception on the intervention by a post-intervention survey consisted of closed-ended and open-ended questions.

   All students who have enrolled in the geriatric course during the study period are invited to participate in this study. A sample size of 85 on each group is expected to provide 90% power to detect difference between sample mean and expected population mean of 0.5, at a significance level of 0.05 (Chow, Shao, & Wang, 2003). Allowing for 10% of attrition, the total number of participants required for this study will be 188. The sample size calculation is estimated from a sample size calculator https://www2.ccrb.cuhk.edu.hk/stat/mean/osm_equality.htm The second part of study is a qualitative descriptive approach to assess on students' perception, attitude and understanding towards elderly patients and their caregivers after YouTube video activities. Approximately 30 students from the intervention group will be invited for focus group discussion till data saturation.
2. Intervention Students of the intervention group are instructed using You Tube video. A series of YouTube video activities is designed to impact students' attitude and understanding on elderly people and their caregivers, fostering them an empathetic attitude towards geriatric clients. The YouTube learning activities will be conducted during tutorial sessions, which consist of five topics, including: elder abuse, elderly poverty, sexuality in elderly people, end-of-life care and successful aging. In each tutorial session, students are required to view a You Tube video clip focusing on weekly learning objectives of the subject. Then, they will be divided into a group of four to six for group discussion on a set of related guiding questions to facilitate their thinking about the elderly clients and their caregivers' situation and their coping strategies.

   Students of the control group are taught with the same content through the usual lecture-based method, without You Tube video.
3. Data analysis The IBM SPSS Version 23.0 (IBM Crop. Armonk, N.Y.) or the latest version, will be used for quantitative data entry and analysis. All statistical tests involved are 2-tailed and the level of significance is set at P ≤ 0.05. Descriptive statistics, will be used to summarize, and present the sample characteristics of the demographic data, survey result and C-JSE-HPS scores. Chi-square Fisher's exact and independent t-tests will be used as appropriate, to assess for homogeneity of the intervention and control groups. The pre-to-post changes of the C-JSE-HPS score among students of intervention and control group will be assessed by using repeated measure ANOVA.

   For focus group interviews, the interview tapes will be transcribed verbatim and field notes will be taken. Data analysis software NVivo 11 or the latest version (QSR International Pty Ltd, Victoria, Australia) that will have used to organize data. Then, the content analysis technique will be adopted, through grouping common sub-themes into themes or nodes, to analysis interview data independently according to the interview guide, with cross-checking for consistency.
4. Ethical consideration Ethical approval of the study was obtained from the Research Ethics Sub-Committee (RESC), Tung Wah College.The purpose, benefits, risk, and procedures of the study was fully explained to the participants and written in the information sheet was issued. Written consent were obtained from study participants before their participation in the study. Participants were informed that they had the right to refuse to respond any questions and withdraw from this study anytime without penalty of any kind. Confidentiality and anonymous of participants were strictly ensured. Permission of interviews to be audio-recorded had been obtained before the focus group interviews.

ELIGIBILITY:
Inclusion Criteria:

* All nursing students of a tertitery institute (the study venue) who had enrolled in the geriatric course at two consecutive semesters during the study period were invited to participate in this study.

Exclusion Criteria:

* Nil

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
The Chinese version of Jefferson Scale of Empathy - Health Professions Students (C-JSE-HPS) | The outcome assessment was taken at baseline, 1 week before study intervention (T0), and (T1)then 1 week after the study intervention, spanned for about 15 weeks
  The Jefferson Scale of Empathy-Health Profession Student Version (JSE-HPS) (Fields et al., 2011) was firstly developed from the original Jefferson Scale of Empathy (Hojat, Gonnella, & Maxwell, 2009). The Taiwan version was translated and validated in 2012. It has been demonstrated with satisfactory psychometric properties, for which the Cronbach's alpha coefficient and the test-retest reliability was 0.93 and 0.92 respectively (Hsaio et al., 2013). It is a 20-items questionnaire, scoring on a 7-point Likert scale ranging from 1= strongly disagree to 7 =strongly agree. 10 out of 20 items in this scale are negatively worded and reversely coded. The JSE-HPS scores range from 20 - 140. Higher scores on the scale reflect for higher level of empathy.
  The study assessed the pre-to-post changes of the C-JSE-HPS score among students of intervention and control group.
Survey on student's perception of the value of YouTube video activities. | The outcome assessment was done at one time point, at 1 week after the study period
  A self-report survey was used to explore student's accessibility to internet and perception of using YouTube as a supplementary learning activity in the intervention group
Focus group interview | Six focus group interviews were conducted after the study intervention, spanned for 4 weeks.
  The focus group interview was a type of semi-structured mode with interview guide, and open-ended format interview. Focus group discussion usually had 6 -12 participants.
  A interview guide was developed by investigators to assess the students of the intervention group, on their perception, attitude and understanding towards elderly patients and their perspectives of elderly care after using YouTube personal stories as a teaching tools in a geriatric course.
  Students of the intervention group would be invited to join for focus group interview for one time after completion of study intervention

CONTACTS AND LOCATIONS:
Overall Officials: Mei Yi Siu, Doctoral, Principal Investigator — Tung Wah College
Locations (1):
- Tung Wah College, Hong Kong, Hong Kong SAR, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The supporting information (as listed above) will become available starting from 1 year after publication for 6 months
Access Criteria: The datasets used and/or analyzed during the current study are available from the corresponding author ( Name: Siu Mei Yi at minniemysiu@gmail.com) on reasonable request. All data analyzed during this study are included in this published article and its supplementary information files.